CLINICAL TRIAL: NCT07166575
Title: Ultrasonographic Assessment of Upper Trapezius Mmorphological Changes in Oral Cancer Patients With Scapular Dyskinesis: An Observational Study
Brief Title: Morphological Changes of Upper Trapezius Muscle After Physotherapy in Oral Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202508084RINA
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Oral Cancer
Keywords: Ultrasonography; Upper Trapezius; Shoulder; Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: B-mode ultrasonography — Thickness and cross-sectional area of upper trapezius muscle

SUMMARY:
The study aims to evaluate the morphological changes of upper trapezius muscle, using B-mode ultrasonography, in patients with oral cancer undergone neck dissection and physiotherapy. It also investigates the relationship between morphological changes and shoulder active range of motion in abduction. Furthermore , the study assesses the potential of B-mode ultrasonography as an objective tool for monitoring outcomes of the rehabilitation in this population.

DETAILED DESCRIPTION:
The study aims to investigate the effect of 8-week physiotherapy on morphological change of upper trapezius muscle in oral cancer patients who have undergone neck dissection. Key outcome measurements include the muscle's thickness and cross-sectional area (CSA), measured via B-mode ultrasonography, as well as the active range of motion (AROM) in shoulder abduction. Neck dissections may result in spinal accessory nerve (CN XI) injury, often leading to shoulder pain, upper trapezius weakness and impaired shoulder mobility. Therefore, understanding the relationship between muscle thickness, CSA, and AROM is important. The study's goal is to explore the correlation between muscle morphological changes and functional outcomes, and further evaluate the role of B-mode ultrasonography as a non-invasive tool in monitoring muscle morphology in shoulder rehabilitation progress with post-surgical oral cancer patients with shoulder dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed oral cancer patients with scapular dyskinesis, who have undergone neck dissections within 3 months
* Able to cooperate with assessments and physical therapy, and capable of understanding and signing the informed consent form.
* Age between 20 and 65 years.

Exclusion Criteria:

* Unable to effectively communicate.
* Diagnosed with conditions affecting motor function.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 10 newly diagnosed oral cancer patients who received neck dissection with scapular dyskinesis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area of upper trapezius muscle | Pre-intervention, 8 weeks post-intervention
  CSA of the upper trapezius muscle is measured via B-mode panoramic ultrasonography. Panoramic B-mode ultrasonography will be performed by placing the probe at the spinous process of the fourth cervical vertebra (C4) and moving it laterally toward the posterior margin of the sternocleidomastoid muscle.
Thickness of upper trapezius muscle | Pre-intervention, 8 weeks post-intervention
  Thickness of upper trapezius muscle is measured via B-mode ultrasonography. The ultrasound probe will be positioned at the midpoint between the spinous process of the seventh cervical vertebra (C7) and the acromion, aligned parallel to the muscle fibers.
Active range of motion in shoulder abduction | Pre-intervention, 8 weeks post-intervention
  AROM in shoulder abduction is measured by a goniometer, with the fulcrum positioned over the anterior aspect of the acromial process. The proximal arm is aligned parallel to the midline of the anterior aspect of the sternum, while the distal arm is aligned with the anterior midline of the humerus.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — National Taiwan University, College of Medicine

REFERENCES:
- [Background] Carenfelt C, Eliasson K. Occurrence, duration and prognosis of unexpected accessory nerve paresis in radical neck dissection. Acta Otolaryngol. 1980 Nov-Dec;90(5-6):470-3. doi: 10.3109/00016488009131750. PMID 7211339
- [Background] Warnakulasuriya S. Global epidemiology of oral and oropharyngeal cancer. Oral Oncol. 2009 Apr-May;45(4-5):309-16. doi: 10.1016/j.oraloncology.2008.06.002. Epub 2008 Sep 18. PMID 18804401
- [Background] van Wilgen CP, Dijkstra PU, van der Laan BF, Plukker JT, Roodenburg JL. Shoulder complaints after neck dissection; is the spinal accessory nerve involved? Br J Oral Maxillofac Surg. 2003 Feb;41(1):7-11. doi: 10.1016/s0266-4356(02)00288-7. PMID 12576033
- [Background] Adigozali H, Shadmehr A, Ebrahimi E, Rezasoltani A, Naderi F. Ultrasonography for the assessment of the upper trapezius properties in healthy females: a reliability study. Muscles Ligaments Tendons J. 2016 May 19;6(1):167-72. doi: 10.11138/mltj/2016.6.1.167. eCollection 2016 Jan-Mar. PMID 27331047
- [Background] Valera-Calero JA, Gallego-Sendarrubias G, Fernandez-de-Las-Penas C, Cleland JA, Ortega-Santiago R, Arias-Buria JL. Cross-sectional area of the cervical extensors assessed with panoramic ultrasound imaging: Preliminary data in healthy people. Musculoskelet Sci Pract. 2020 Dec;50:102257. doi: 10.1016/j.msksp.2020.102257. Epub 2020 Sep 11. PMID 32947195